CLINICAL TRIAL: NCT02692105
Title: A Phase III Randomized Pilot Study of Low Dose Rate Compared to High Dose Rate Prostate Brachytherapy for Favourable Risk and Low Tier Intermediate Risk Prostate Cancer
Brief Title: Comparison of HDR vs. LDR Brachytherapy as Monotherapy for Intermediate Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Juanita Crook, Professor of Radiation Oncology, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H15-02103
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: prostate adenocarcinoma; intermediate risk group; brachytherapy; High Dose Rate vs Low Dose Rate; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose rate brachytherapy (Active Comparator): Device: Radiation Low dose rate prostate brachytherapy is delivered under anaesthesia in a single 1.5-2 hour procedure as an out-patient. The men return 4 weeks later for detailed imaging to assess implant quality.
  Interventions: Radiation: Low dose rate prostate brachytherapy
- High dose rate brachytherapy (Experimental): Device: Radiation High dose rate prostate brachytherapy is delivered in 2 procedures, 2 weeks apart, also under anaesthesia, but no follow-up imaging visit is required.
  HDR brachytherapy is also accomplished as an out-patient.
  Interventions: Radiation: High Dose Rate prostate brachytherapy

INTERVENTIONS:
Radiation: Low dose rate prostate brachytherapy — Permanent implantation of radioactive Iodine-125 seeds under anesthesia with ultrasound guidance
  Other Names: LDR brachytherapy, seed brachytherapy
  Arms: Low dose rate brachytherapy
Radiation: High Dose Rate prostate brachytherapy — Temporary implantation of radioactive material into the prostate in the form of a stepping source of Iridium 192 that travels through 16-18 needles or catheters strategically placed through the prostate
  Other Names: HDR brachytherapy
  Arms: High dose rate brachytherapy

SUMMARY:
This study will offer men with intermediate risk prostate cancer who are suitable for, and interested in, prostate brachytherapy, the opportunity to be randomized between low dose rate (LDR) brachytherapy using permanent implantation of radioactive seeds (the current standard of care in BC) and high dose rate (HDR) or temporary brachytherapy which is also available as a standard of care in BC but only when used as a boost in addition with external beam radiotherapy. In addition, men will be offered the opportunity for testing the aggressiveness of their cancer using Cell Cycle Progression Gene Profile.

DETAILED DESCRIPTION:
Purpose:

To conduct a Phase III randomized trial for favorable tier intermediate risk prostate cancer and selected favorable risk tumors to evaluate the difference in Quality of Life in the urinary domain between LDR and HDR brachytherapy.

Hypothesis:

Because of more rapid dose delivery with HDR compared to LDR brachytherapy (15 minutes vs. 6 months) and more precise control of dose to adjacent critical structures (prostatic and bulbo-membranous urethra and anterior rectal wall), HDR prostate brachytherapy has been associated with more rapid recovery from acute symptoms and a more favorable side effect protocol when used as a boost in combination with external beam radiotherapy. The hypothesis is that this advantage will be maintained when brachytherapy is used as monotherapy without the addition of external beam radiation.

Justification:

In British Columbia, LDR prostate brachytherapy is the current standard for selected men with favorable risk prostate cancer who are not suitable for, or willing to accept active surveillance, and for men with favorable intermediate risk prostate cancer. LDR brachytherapy has been available in BC for over 15 years and is highly effective with 7-year biochemical disease-free rates of ~95%. However, this type of treatment has a prolonged recovery phase with return to baseline urinary function taking 6 to 12 months. This is partly due to the fact that the radiation is delivered over a 6 month period from the implanted seeds, and partly due to uncertainty in final seed placement. HDR brachytherapy has the advantage of delivering treatment very rapidly over 15-20 minutes, and also exploits the radiobiologic nature of prostate cancer which is more responsive to large doses of radiotherapy. Experience with using HDR brachytherapy as a boost has shown a much reduced impact on quality of life.

Objectives:

Primary: To evaluate the difference in QOL in the urinary domain between LDR and HDR brachytherapy using the urinary domain of the EPIC prostate cancer specific QOL questionnaire.

Secondary:

* To assess differences in the bowel and sexual domains of the EPIC prostate cancer specific QOL questionnaire between the 2 treatments
* To asses time to recovery of the IPS Score which is widely used to assess urinary function after prostate cancer treatment. The time to return to baseline +/- 3 points will be determined.
* Acute and long-term toxicity will be graded using the Common Terminology Criteria for Adverse Events (CTCAE V4) at each follow up time point
* TRUS- MRI fusion will be developed within our planning software to facilitate treatment planning
* To assess treatment efficacy, PSA will be recorded every 6 months to 5 years and then annually to 10 years and prostate re-biopsy will be performed at 36 months after radiotherapy.

Optional:

For those patients consenting to targeted biopsies under anaesthesia at the start of their brachytherapy procedure (separate consent)

* Verify MRI-TRUS fusion accuracy
* Correlate Cell Cycle Progression scores with outcome.

Research Method:

Multiparametric MRI (mpMRI)will be performed on all men as a staging procedure to ensure appropriateness for brachytherapy as monotherapy (without the addition of external beam radiotherapy or hormone therapy). The value of mpMRI in staging prostate cancer is widely recognized. Previous studies have shown that over 90% of intermediate risk cancers are visible on mpMRI. The MR images will be fused with the planning trans rectal ultrasound (TRUS) for each patient, ensuring adequate dose coverage of the lesion.

For those patients consenting to optional biopsies under anesthesia, accuracy of the fusion will be verified by obtaining 2 biopsies of the visualized lesion under TRUS guidance at the start of the brachytherapy procedure.

Follow up is as per standard practice to assess urinary, bowel and sexual side effects. In addition to the standard forms, patients will also complete an EPIC questionnaire. The questionnaires are completed every 3 months for 1 year and then every 6 months to 3 years and then annually, as per the standard follow up schedule.

Once the biopsy material has been pathologically confirmed to contain the target lesion, the aggressiveness will be assessed through Cell Cycle Progression (CCP) Gene Profile testing.

Men may be randomized to the type of brachytherapy and decline the biopsies. This initial protocol is a Pilot that will test feasibility of the randomization (patient acceptance). The aim is to accrue 60 men over 18-24 months and if achieved then apply to expand to a total of 200 men.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage T1c-T2b, PSA < 20, Gleason < 8
* ECOG 0-1
* Low tier intermediate-risk prostate cancer is defined by;

  o a single NCCN intermediate risk factor (either Gleason 7(3+4) and PSA < 10 ng/ml OR Gleason 6 and PSA 10-20 ng/ml)
* Extensive favorable-risk disease is defined as:

  * clinical stage T1c-T2a
  * PSA < 10
  * Gleason 6
  * ≥ 50% of biopsy cores containing cancer
  * PSA density > 0.2 ng/cc
* Selected intermediate risk patients not defined above

  * - T1c/T2a
  * - PSA < 10
  * -Gleason 4+3
  * -< 33% of cores involved
  * -Max tumour length in any core 10 mm
* No androgen deprivation therapy (ADT)
* Prostate volume by TRUS ≤ 60 cc.
* Not eligible for, or accepting of, active surveillance according to NCCN guidelines.
* Signed study specific informed consent.

Exclusion Criteria:

* Prior radical surgery for carcinoma of the prostate,
* Prior pelvic radiation
* Prior chemotherapy for prostate cancer,
* Prior TURP or cryosurgery of the prostate
* Claustrophobic or unable to undergo MRI

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The difference in Quality of Life in the urinary domain between LDR and HDR brachytherapy. | 0-36 months
  The urinary domain of the EPIC prostate cancer specific QOL questionnaire will be assessed.

SECONDARY OUTCOMES:
Quality of Life in the bowel and sexual domains | 0-36 months
  The EPIC score in the bowel and sexual domains will be evaluated at baseline, 1, 3, 6, 12, 24 and 36 months
Time to return to baseline +/- 3 points for the International Prostate Symptom Score | 0-36 months
  The IPS Score will be assessed at baseline, 1, 3, 6, 12, 24 and 36 months
Acute and long term toxicity | 0-10 years
  Acute and long-term toxicity will be graded using the Common Terminology Criteria for Adverse Events (CTCAE V4) at each follow up time point
TRUS- MRI fusion | baseline
  TRUS- MRI fusion will be developed within our planning software to facilitate treatment planning
Biochemical Outcome | 5-10 years
  PSA will be recorded every 6 months to 5 years and then annually to 10 years
Histologic Outcome | 3 years
  Prostate re-biopsy will be performed at 36 months to assess the local efficacy of treatment
Cell cycle progression score | one month
  For those patients consenting to targeted biopsies under anesthesia at the start of their brachytherapy procedure (separate optional consent) MRI-TRUS fusion accuracy will be verified by targeted biopsies and Biopsy material will be sent for genetic testing to determine Cell cycle Progression scores for both arms of the trial to ultimately correlate with outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Halperin, MD, Study Director — British Columbia Cancer Agency Program Director
Locations (1):
- British Columbia Cancer Agency Center for the Southern Interior, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crook J, Ots A, Gaztanaga M, Schmid M, Araujo C, Hilts M, Batchelar D, Parker B, Bachand F, Milette MP. Ultrasound-planned high-dose-rate prostate brachytherapy: dose painting to the dominant intraprostatic lesion. Brachytherapy. 2014 Sep-Oct;13(5):433-41. doi: 10.1016/j.brachy.2014.05.006. Epub 2014 Jun 20. PMID 24958556
- [Background] Batchelar D, Gaztanaga M, Schmid M, Araujo C, Bachand F, Crook J. Validation study of ultrasound-based high-dose-rate prostate brachytherapy planning compared with CT-based planning. Brachytherapy. 2014 Jan-Feb;13(1):75-9. doi: 10.1016/j.brachy.2013.08.004. Epub 2013 Sep 27. PMID 24080299
- [Background] Schmid M, Crook JM, Batchelar D, Araujo C, Petrik D, Kim D, Halperin R. A phantom study to assess accuracy of needle identification in real-time planning of ultrasound-guided high-dose-rate prostate implants. Brachytherapy. 2013 Jan-Feb;12(1):56-64. doi: 10.1016/j.brachy.2012.03.002. Epub 2012 Apr 17. PMID 22513104